CLINICAL TRIAL: NCT04121078
Title: A Phase 1, Open-Label, Randomized, Two-Way Crossover Study to Evaluate the Effect of Single-Dose Intravenous Rifampin as a Prototypic Inhibitor of OATP1B1 and OATP1B3 on the Single-Dose Pharmacokinetics of Oral TAK-906 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Single-Dose Intravenous Rifampin as a Prototypic Inhibitor of Organic Anion Transporting Polypeptide (OATP) 1B1 and OATP1B3 on the Single-Dose Pharmacokinetics (PK) of Oral TAK-906 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-906-1009; U1111-1240-6352 (Other: WHO)
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — trazpiroben; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB: TAK-906 25 mg + TAK-906 25 mg and Rifampin 600 mg (Experimental): TAK-906 25 milligram (mg) (Treatment A), capsule, orally, once on Day 1 of Study Period 1, followed by a washout period of at least 7 days, further followed by rifampin 600 mg, infusion, once, intravenously over 30 minutes along with TAK-906 25 mg (Treatment B), capsule, orally, once immediately after the end of infusion on Day 1 of Study Period 2.
  Interventions: Drug: TAK-906; Drug: Rifampin
- Sequence BA: TAK-906 25 mg and Rifampin 600 mg + TAK-906 25 mg (Experimental): Rifampin 600 mg, infusion, once, intravenously over 30 minutes along with TAK-906 25 mg (Treatment B), capsule, orally, once immediately after the end of infusion on Day 1 of Study Period 1 followed by a washout period of at least 7 days, further followed by TAK-906 25 mg (Treatment A), capsule, orally, once on Day 1 of Study Period 2.
  Interventions: Drug: TAK-906; Drug: Rifampin

INTERVENTIONS:
Drug: TAK-906 — TAK-906 capsule.
Drug: Rifampin — Rifampin infusion.

SUMMARY:
The purpose of this study is to evaluate the effect of single dose intravenous rifampin on the single-dose PK of orally administered TAK-906.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. TAK-906 is being tested to evaluate the effect of single dose intravenous rifampin on the single-dose PK of oral TAK-906 in healthy adult participants.

The study will enroll approximately 12 participants. Participants will be randomly assigned to one of the two treatment sequences AB or BA:

* Sequence AB: TAK-906 25 mg, followed by a washout period of at least 7 days, then Rifampin 600 mg and TAK-906 25 mg
* Sequence BA: Rifampin 600 mg and TAK-906 25 mg, followed by a washout period of at least 7 days, then TAK-906 25 mg

This single center trial will be conducted in the United States. The overall time to participate in this study is 49 Days. All participants will make final visit 14 days after receiving their last dose of study drug for follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dosing and throughout the study, based on screening urine cotinine test.
2. Body Mass Index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 30.0 kilogram per square meter (kg/ m^2) at screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the investigator or designee.

Exclusion Criteria:

1. Positive urine drug or alcohol results at screening and each check in.
2. Positive urine cotinine at screening.
3. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
4. QT interval with Fridericia's correction (QTcF) interval is >450 millisecond (msec) or ECG findings are deemed abnormal with clinical significance by the investigator or designee at screening.
5. Estimated creatinine clearance <90 milliliter per minute (mL/min) at screening.
6. Has been on a diet incompatible with the on-study diet, in the opinion of the investigator or designee, within the 30 days prior to the first dosing and throughout the study.
7. Donation of blood or significant blood loss (example, approximately 500 milliliter [mL]) within 56 days prior to the first dosing.
8. Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Mukker JK, Dukes G, Tolkoff M, Wang L, Almansa C, Huh SY, Nishihara M, Ramsden D, Chen C. The pharmacokinetics of oral trazpiroben (TAK-906) after organic anion transporting polypeptide 1B1/1B3 inhibition: A phase I, randomized study. Clin Transl Sci. 2022 Jun;15(6):1532-1543. doi: 10.1111/cts.13274. Epub 2022 May 5. PMID 35460165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 15 October 2019 to 16 November 2019.
Pre-assignment Details: Healthy participants were enrolled in 1 of the 2 treatment sequences of this 2-period crossover study to receive TAK-906 25 milligram (mg) alone (Treatment A) and TAK-906 25 mg along with rifampin 600 mg (Treatment B).
Groups:
- Sequence AB: TAK-906 25 mg + TAK-906 25 mg and Rifampin 600 mg: TAK-906 25 mg (Treatment A), capsule, orally, once on Day 1 of Study Period 1, followed by a washout period of at least 7 days, further followed by rifampin 600 mg, infusion, intravenously along with TAK-906 25 mg (Treatment B), capsule, orally, once immediately after the end of infusion on Day 1 of Study Period 2.
- Sequence BA: TAK-906 25 mg and Rifampin 600 mg + TAK-906 25 mg: Rifampin 600 mg, infusion, intravenously along with TAK-906 25 mg (Treatment B), capsule, orally, once immediately after the end of infusion on Day 1 of Study Period 1, followed by a washout period of at least 7 days, further followed by TAK-906 25 mg (Treatment A), capsule, orally, once on Day 1 of Study Period 2.
Period: Study Period 1 (1 Day)
Arm/Group | Sequence AB: TAK-906 25 mg + TAK-906 25 mg and Rifampin 600 mg | Sequence BA: TAK-906 25 mg and Rifampin 600 mg + TAK-906 25 mg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | Sequence AB: TAK-906 25 mg + TAK-906 25 mg and Rifampin 600 mg | Sequence BA: TAK-906 25 mg and Rifampin 600 mg + TAK-906 25 mg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Study Period 2 (1 Day)
Arm/Group | Sequence AB: TAK-906 25 mg + TAK-906 25 mg and Rifampin 600 mg | Sequence BA: TAK-906 25 mg and Rifampin 600 mg + TAK-906 25 mg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence AB: TAK-906 25 mg + TAK-906 25 mg and Rifampin 600 mg | Sequence BA: TAK-906 25 mg and Rifampin 600 mg + TAK-906 25 mg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (13.47) | 38.0 (8.12) | 37.3 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  Black or African American, White | 1 | 0 | 1
  White | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 74.73 (9.943) | 84.25 (13.581) | 79.49 (12.389)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.3 (11.74) | 177.0 (9.38) | 174.7 (10.42)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m˄2)] | 25.168 (2.3720) | 26.770 (1.8285) | 25.969 (2.1856)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-906
Time Frame: Day 1: time zero and at multiple time points (up to 48 hours) post dose
Population: The pharmacokinetic (PK) set consisted of all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A: TAK-906 25 mg: TAK-906 25 mg, capsule, orally, once on Day 1 of either Study Period 1 or 2.
- Treatment B: Rifampin 600 mg and TAK-906 25 mg: Rifampin 600 mg, infusion, intravenously along with TAK-906 25 mg, capsule, orally, once immediately after the end of infusion on Day 1 of either Study Period 1 or 2.
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 14.37 (38.7) | 89.62 (68.6)
Statistical Analysis 1: Comparison: Treatment A: TAK-906 25 mg vs Treatment B: Rifampin 600 mg and TAK-906 25 mg; Test type: Equivalence — Point estimate and its 90% confidence interval (CI) were calculated for Treatment B to Treatment A ratio of geometric means for Cmax based on the mixed-effect model of log-transformed Cmax with sequence, treatment, and period as fixed effects, and participant nested within sequence as a random effect. Bioequivalence was concluded if the 90% CI for the ratio of geometric means is entirely contained within 80% to 125% for Cmax. No adjustments were made for multiplicity; Geometric Mean Ratio = 6.24, 90% CI 2-sided [4.62 to 8.42]

2. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-906
Time Frame: Day 1: time zero and at multiple time points (up to 48 hours) post dose
Population: The PK set consisted of all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 32.68 (23.9) | 168.5 (49.9)
Statistical Analysis 1: Comparison: Treatment A: TAK-906 25 mg vs Treatment B: Rifampin 600 mg and TAK-906 25 mg; Test type: Equivalence — Point estimate and its 90% CI were calculated for Treatment B to Treatment A ratio of geometric means for AUC∞ based on the mixed-effect model of log-transformed AUC∞ with sequence, treatment, and period as fixed effects, and participant nested within sequence as a random effect. Bioequivalence was concluded if the 90% CI for the ratio of geometric means is entirely contained within 80% to 125% for AUC∞. No adjustments were made for multiplicity; Geometric Mean Ratio = 5.16, 90% CI 2-sided [4.25 to 6.25]

3. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-906
Time Frame: Day 1: time zero and at multiple time points (up to 48 hours) post dose
Population: The PK set consisted of all participants who received study drug and had at least 1 measurable plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 32.32 (23.8) | 168.3 (49.9)
Statistical Analysis 1: Comparison: Treatment A: TAK-906 25 mg vs Treatment B: Rifampin 600 mg and TAK-906 25 mg; Test type: Equivalence — Point estimate and its 90% CI were calculated for Treatment B to Treatment A ratio of geometric means for AUClast based on the mixed-effect model of log-transformed AUClast with sequence, treatment, and period as fixed effects, and participant nested within sequence as a random effect. Bioequivalence was concluded if the 90% CI for the ratio of geometric means is entirely contained within 80% to 125% for AUClast. No adjustments were made for multiplicity; Geometric Mean Ratio = 5.21, 90% CI 2-sided [4.29 to 6.32]

4. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 14 days after the last dose of study drug in Study Period 2 (up to Day 23)
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
Participants | 6 | 2

5. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign Values
Time Frame: Baseline up to 14 days after the last dose of study drug in Study Period 2 (up to Day 23)
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Time Frame: Baseline up to 14 days after the last dose of study drug in Study Period 2 (up to Day 23)
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Values
Time Frame: Baseline up to 14 days after the last dose of study drug in Study Period 2 (up to Day 23)
Population: The safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events (AEs) that started after the first dose of study drug and no more than 14 days after the last dose of study drug in Study Period 2 (up to Day 23)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Treatment A: TAK-906 25 mg | Treatment B: Rifampin 600 mg and TAK-906 25 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: TAK-906 25 mg (N=12) | Treatment B: Rifampin 600 mg and TAK-906 25 mg (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT04121078/SAP_000.pdf
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT04121078/Prot_001.pdf